CLINICAL TRIAL: NCT06967233
Title: Analysis of the Current Situation of Diagnosis and Treatment of Pancreatic Cancer: Multimodal Managements for Metastatic Pancreatic Cancer
Brief Title: Multimodal Managements for Metastatic Pancreatic Cancer.
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Other Study IDs: Multimodal-MPC
Record Dates: First submitted 2025-05-02; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Combined Modality Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multimodal treatment — Surgical resection, locoregional liver-directed treatments and continuous systemic treatment in patients with liver metastatic pancreatic cancer

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) remains a challenging malignancy, with over 300,000 patients diagnosed annually worldwide. Patients with metastatic pancreatic cancer (MPC) are generally not considered appropriate for operative management because it would not improve their prognosis.

Developments in modern surgery and systemic treatment over the past decade have substantially improved the oncological outcomes for patients with PDAC. The prognosis can be further improved by using novel combined regimens. Systemic treatment is advantageous as it allows biological selection of patients and control of systemic lesions in patients with PDAC with only hepatic metastases (Hep-MPC), which may increase the likelihood of radical tumor resection and improved survival. Therefore, there is a strong need to reassess the value of surgery in Hep-MPC.

Locoregional liver-directed treatments (LLDTs) are safe and efficient methodologies and have thus become the standard of care for patients with metastatic colorectal cancer (MCC) with liver-only or liver-dominant metastases. LLDT therapies include local liver resection, radiofrequency ablation (RFA), hepatic artery infusion pump chemotherapy (HAIP), stereotactic body radiation therapy (SBRT), and selective internal radiation therapy with yttrium-90 embolization (Y90). These therapies have been reported to influence the overall survival (OS), progression-free survival (PFS), and conversion to resection in patients with metastatic colorectal cancer. However, the data on the survival outcomes of conversion surgery and the clinical application of LLDT in Hep-MPC are sparse. Therefore, it remains unclear what types of treatment, based on the survival benefit, might actually be the optimal approach for Hep-MPC after effective systemic treatment.

The present study aims to clarify the selection criteria of conversion surgery for Hep-MPC and explore the prognostic significance for its multimodal management, including surgical resection and/or LLDT.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years (at diagnosis).
* Cytologically or histologically confirmed pancreatic adenocarcinoma.
* Synchronous liver metastatic disease (at diagnosis).
* No evidence of extrahepatic metastases (at diagnosis.)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
* Eligible for multimodal treatment.

Exclusion Criteria:

* Multi-organ metastatic pancreatic cancer.
* Contraindications to surgical resection or systemic treatment.
* Inability to participate in follow-up assessments.
* History of other malignancies.
* Refusal of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were cytologically or histologically diagnosed with pancreatic cancer, as well as with the primary tumor and liver metastasis. The primary and metastatic lesions were determined using CT and MRI.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | From the date of treatment initiation to the date of death or the last date of follow-up (up to 60 months)
  Calculated from the date of treatment initiation to the date of death or the last date of follow-up

SECONDARY OUTCOMES:
Progression free survival | From the date of treatment initiation to the date of disease progression or death, whichever occurred first (up to 60 months).
  The duration between the date of treatment initiation and disease progression or death, whichever occurred first.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital, Zhejiang university school of medicine, Hangzhou, Zhejiang, China